CLINICAL TRIAL: NCT00537212
Title: A Single-Center, Prospective, Single-Blinded, Pilot Study to Compare the Effect of Diet in Overweight or Obese Patients With Psoriasis on Light Therapy
Brief Title: Study of the Effect of Diet in Overweight or Obese Patients With Psoriasis on Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagel, Jerry, M.D. (Individual)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jerry Bagel MD, Director, Bagel, Jerry, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0-001
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis; Weight Loss; Diet
Keywords: Psoriasis; Weight loss; diet
MeSH Terms: conditions — Psoriasis; Weight Loss | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Subjects will receive phototherapy and dietary counselling consistent with "The South Beach diet."
  Interventions: Other: The South Beach Diet
- 2 (Active Comparator): Subjects will receive phototherapy and dietary counselling consistent with "The Ornish Diet."
  Interventions: Other: The Ornish Diet
- 3 (Sham Comparator): Subjects will receive phototherapy alone, without dietary counselling.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: The South Beach Diet — Subjects will receive dietary counselling aimed at reducing simple carbohydrates and increasing weight loss. Subjects also receive a copy of "The South Beach Diet."
  Arms: 1
Other: The Ornish Diet — Subjects will receive dietary counselling aimed to reduce fat consumption and increase weight loss. Subjects also receive a copy of "The Ornish Diet" book.
  Arms: 2
Other: Control Group — This group will receive phototherapy alone. They will not be counselled or give literature on a particular diet.
  Other Names: Phototherapy only
  Arms: 3

SUMMARY:
The association between psoriasis and obesity has been questioned by physicians for many years. Studies have shown that the risk of having psoriasis is increased in people with a high body mass index, which is a measurement of obesity. There have been case reports of remission of psoriasis after gastric bypass surgery. Furthermore, other studies have shown that certain inflammatory diseases (such as rheumatoid arthritis) can be improved by dietary changes. The purpose of this study is to assess whether a low carbohydrate or low fat diet can be helpful in the treatment of psoriasis.

DETAILED DESCRIPTION:
This study involves the use of diet as a therapeutic agent in subjects with obesity and psoriasis who are eligible for and willing to undergo phototherapy. Subjects undergoing phototherapy alone will be compared to subjects randomized to receive phototherapy and dietary modification with the goal of weight loss. The primary objective is to determine the success rate of weight loss programs in the setting of psoriasis. Secondary objectives include evaluating the effect of weight loss on efficacy of narrow band ultraviolet B phototherapy, and assessing the efficacy of lower carbohydrate and low fat diets in psoriatic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18
2. PASI score greater than 10
3. BMI greater than 25
4. Subjects must be willing and eligible to undergo phototherapy and
5. Willing to stop all other psoriasis therapies

Exclusion Criteria:

1. History of failure to respond to NB-UVB in the past.
2. Presence of predominantly guttate, erythrodermic, or pustular psoriasis or any skin condition that would interfere with evaluation of effect of study. intervention .
3. Treatment with systemic antibiotics, topical steroids (except to groin and face), topical Vitamin A or D analogs, or ultraviolet B therapy within 2 weeks of study initiation.
4. Use or oral or parenteral corticosteroids.
5. Use of appetite suppressants or other medications know to affect appetite or weight.
6. Treatment with biologic therapy in the past 3 months.
7. History of cutaneous malignancy, including any squamous cell carcinoma or melanoma or more than two basal cell carcinomas, current actinic keratoses or atypical moles.
8. Evidence of photosensitivity disorder (e.g.polymorphous light eruption.
9. Use of other investigational drugs, any systemic psoriasis therapy, psoralen plus ultraviolet A therapy (PUVA) within 4 weeks of study drug initiation.
10. Subjects who are currently achieving good clinical control of their psoriasis on their current therapy.
11. Concomitant serious illness or medical condition that may interfere with participation in the study including renal failure, hepatic failure or systemic lupus erythematosus.
12. Subject currently enrolled in another investigational device or drug trial(s), or that may compromise the safety of data collection.
13. Any condition judged by the investigator to cause this clinical trial to be detrimental to the patient.
14. Subject known to be pregnant or breastfeeding.
15. Evidence of skin conditions (e.g.,eczema) other than psoriasis that would interfere with study-related evaluations of psoriasis.
16. History of psychiatric disease that would interfere with the patient's ability to comply with the study protocol.
17. History of non-compliance with other therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PASI improvement | 12 weeks

SECONDARY OUTCOMES:
which group's PASI did better | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, M.D., Principal Investigator — Psoriasis Treatment Center of Central New Jersey
Locations (1):
- Jerry Bagel, East Windsor, New Jersey, United States